CLINICAL TRIAL: NCT01497028
Title: Prospective Randomized Clinical Trial of Plicated Laparoscopic Adjustable Gastric Banding
Brief Title: Plicated Laparoscopic Adjustable Gastric Banding (Lap Band)
Status: Terminated | Type: Observational
Sponsor: Jacksonville Surgical Associates (Other)
Responsible Party: Principal Investigator, Robert Cywes, M.D., PhD, Prinicipal Investigator, Jacksonville Surgical Associates
Other Study IDs: PLAGB
Record Dates: First submitted 2011-11-22; First posted 2011-12-22 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2011-12

CONDITIONS: Weight Loss
Keywords: Co-morbid disease resolution
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Plicated Gastric Banding
  Interventions: Procedure: PLAGB will be studied and compared to the standard LAGB procedure through a dual center, prospective clinical trial.
- Standard Gastric Banding
  Interventions: Procedure: PLAGB will be studied and compared to the standard LAGB procedure through a dual center, prospective clinical trial.

INTERVENTIONS:
Procedure: PLAGB will be studied and compared to the standard LAGB procedure through a dual center, prospective clinical trial. — PLAGB will be studied and compared to the standard LAGB procedure through a dual center, prospective clinical trial.

SUMMARY:
This is a dual site, prospective study which will compare plicated-Laparoscopic Adjustable Gastric Banding (PLAGB) to standard LABG (SLAGB) to identify significant differences in bariatric surgical outcomes

* Weight Loss
* Co-morbid disease resolution

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following criteria to be eligible for study entry:

* Age between 18 - 80 years, and
* Severely or Morbidly obese:

  * BMI > 35, or
  * BMI > 30 + co-morbid obesity related disease condition
* Without any contraindications to bariatric surgery, and
* Without any metabolic or medically correctable causes for obesity (eg. Untreated hypothyroidism, Prader-Willi, etc.)
* Patients who have had previous LAGB surgery requiring revision for complications such as slippage, stalled weight loss or weight regain

Exclusion Criteria:

Subjects meeting the following criteria will be excluded from study entry:

* Any patient not meeting the inclusion criteria
* Patients with any major medical problems contraindicating surgery
* Patients with a medically treatable cause of obesity (eg. untreated hypothyroidism, Prader-Willi, etc.)
* Patients who elect to undergo a surgery other than a PLAGB or SLAGB
* Pregnant or planning pregnancy within 12 months
* Alcohol or drug addiction
* Established infection anywhere in the body at the time of surgery
* Previous history of other bariatric surgery (except LAGB)
* Family or patient history of autoimmune disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients between the ages of 18-80 years of age who are severly or morbidly obese and meet NIH and FDA criteria for baratric surgery (BMI>30+ co-morbid disease or BMI>35) who are undergoing baratric surgery at Jacksonville Surgical Associates, P.A. or Ventura Advanced Surgical Associates will be returned. All enrolled patients will be assigned to either the SLAGB (control)group or the PLAGB (study) group.
Sampling Method: Probability Sample
Dates: Start 2011-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Ventura Advanced Surgical Associates, Ventura, California
  - Jacksonville Surgical Associates, Jacksonville, Florida